CLINICAL TRIAL: NCT06525311
Title: A Phase 1 Open-Label Study to Evaluate the Pharmacokinetics and Safety of K-808 (Pemafibrate) in Subjects With Primary Biliary Cholangitis With Compensated Cirrhosis and Without Cirrhosis
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of K-808 (Pemafibrate) in Subjects With Primary Biliary Cholangitis With Compensated Cirrhosis and Without Cirrhosis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K-808-1.01
Record Dates: First submitted 2024-06-27; First posted 2024-07-29 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Primary Biliary Cholangitis; Compensated Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PBC w/o CIRR (Experimental): K-808 single dose followed by multiple-dose treatment period.
  Interventions: Drug: K-808
- PBC w/ CIRR CP-A (Experimental): K-808 single dose followed by optional multiple-dose treatment period.
  Interventions: Drug: K-808

INTERVENTIONS:
Drug: K-808 — K-808 single or multi dose extended-release tablets
  Other Names: Pemafibrate

SUMMARY:
A Trial to Investigate the Pharmacokinetics (PK) Effects and Safety Profile of K-808 (Pemafibrate) in Primary Biliary Cholangitis (PBC) Subjects with and without Cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a PBC diagnosis as demonstrated by the presence of ≥2 of the following three diagnostic criteria (Lindor et al, 2019; Hirschfield et al, 2017):

  1. History of ALP above ULN for at least 6 months
  2. History of positive antimitochondrial antibody (AMA) titer or positive PBC-specific antinuclear antibody (ANA) titers
  3. Historical liver biopsy consistent with PBC
* Has PBC with cirrhosis Child-Pugh grade A (well-compensated disease; score 5 to 6) at Screening. Group 2 (PBC w/ CIRR CP-A) only
* Male or female participant is ≥18 years of age at consent.
* Able to understand and comply with study requirements and procedures and provide written informed consent.
* Meet all other inclusion criteria outlined in the clinical study protocol.

Exclusion Criteria:

* Female subject of childbearing potential who is known to be pregnant, has a positive pregnancy test (serum test, or urine test that is confirmed by a positive serum pregnancy test), or is lactating and breastfeeding, or planning to become pregnant or breastfeed during the study.
* Subject has had ongoing conditions that may affect drug absorption such as gastroparesis, intestinal obstruction, severe gastritis, severe gastric reflux syndrome, conditions causing frequent vomiting and/or diarrhea.
* Subject who has participated in another investigational drug, biologic, or medical device study within five half-lives of the agent (or within 8 weeks when half-life is unknown) prior to the first dose of study drug, or prior participation in an investigational antibody drug study within 6 months prior to the first dose of study drug. Participation in noninterventional studies (eg, observational studies, registries) is allowed.
* Meet any other exclusion criteria outlined in the clinical study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
PK parameters after a single dose of K-808: Area under the curve from 0 to infinity (AUC0-inf) | Day 1 - Day 3
PK parameters after a single dose of K-808: Area under the curve from time 0 to last quantifiable time (AUC0-t) | Day 1 to Day 3
PK parameters after a single dose of K-808: Observed maximum plasma concentration (Cmax) | Day 1 to Day 3
PK parameters after a single dose of K-808: Time to reach observed maximum plasma concentration (Tmax) | Day 1 to Day 3
PK parameters after a single dose of K-808: kel | Day 1 to Day 3
PK parameters after a single dose of K-808: Apparent first-order terminal elimination half-life (t½) | Day 1 to Day 3.
PK parameters after a single dose of K-808: Apparent total volume of distribution estimated based on the terminal phase (Vd/F) | Day 1 to Day 3
PK parameters after a single dose of K-808: Apparent plasma clearance after extravascular administration (CL/F) | Day 1 to Day 3
PK parameters after a single dose of K-808: Mean resistance time from time 0 to last measurable concentration (MRT0-t) | Day 1 to Day 3
PK parameters after a single dose of K-808: MRT from time 0 extrapolated to infinity (MRT0-inf) | Day 1 to Day 3
Trough concentrations after multiple dosing of K-808 | Day 4 - Day 6
PK parameters at steady state after multiple dosing of K-808: Area under the curve over the dosing interval (AUC0-tau) | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: Cmax | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: Tmax | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: kel | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: t½ | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: Vd,ss/F at steady state | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: CLss/F at steady state | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: MRT at steady state (MRTss) | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: Observed accumulation ratio based on the AUC (RobsAUC) | Day 6 to Day 8

SECONDARY OUTCOMES:
PK parameters of K-808 metabolites after a single dose: AUC0-inf | Day 1 - Day 3
PK parameters of K-808 metabolites after a single dose: AUC0-t | Day 1 to Day 3
PK parameters of K-808 metabolites after a single dose: Cmax | Day 1 to Day 3
PK parameters of K-808 metabolites after a single dose: Tmax | Day 1 to Day 3
PK parameters of K-808 metabolites after a single dose: kel | Day 1 to Day 3
PK parameters of K-808 metabolites after a single dose: t½ | Day 1 to Day 3
PK parameters of K-808 metabolites after a single dose: MRT0-t | Day 1 to Day 3
PK parameters of K-808 metabolites after a single dose: MRT0-inf | Day 1 to Day 3
PK parameters at steady state after multiple dosing of K-808: AUC0- tau | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: Cmax | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: Tmax | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: kel | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: t½ | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: (MRTss) | Day 6 to Day 8
PK parameters at steady state after multiple dosing of K-808: (RobsAUC) | Day 6 to Day 8
Trough concentrations after multiple dosing of K-808 | Day 4 to Day 6
To assess the safety and tolerability of K-808 | 5 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sara Neville, MD, Study Director — Kowa Research Institute, Inc.
Locations (10):
- United States (6):
  - Arizona Liver Health, Chandler, Arizona
  - Southern California Research Center, Inc, Coronado, California
  - Indiana University School of Medicine - Indianapolis, Indianapolis, Indiana
  - Houston Research Institute, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
- Japan (4):
  - 303, Fukuoka
  - 302, Kita-gun
  - 304, Shinjuku-ku
  - 301, Yufu